CLINICAL TRIAL: NCT03542149
Title: Phase 1b to Assess Safety, Tolerability, Pharmacokinetic Profile, and Antimalarial Activity of Single Doses of Co-administered OZ439and PQP Against Early Plasmodium Falciparum Blood Stage Infection in Healthy Adult Volunteers
Brief Title: Safety, Tolerability and Antimalarial Activity of Single Doses of OZ439 and PQP
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: QIMR Berghofer Medical Research Institute (Other); Clinical Network Services (CNS) Pty Ltd (Industry); Q-Pharm Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: QP17C19
Record Dates: First submitted 2018-05-11; First posted 2018-05-31 (Actual); Results first posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2023-12

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria | interventions — piperaquine; artefenomel

STUDY DESIGN:
Intervention Model Description: Based on safety and tolerability data up to Day 35 post-dose, and pharmacokinetic/pharmacodynamic (PK/PD) analysis outcomes (based on PD data up to Day 35 and PK data up to Day 28 post-dose) of the drugs given in combination, the dose(s) for the subsequent cohort will be determined. A similar analysis will be done at the end of cohort 2 combining cohorts 1 and 2 data to decide the dose(s) to be tested in cohort 3.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP (Experimental): 200mg of OZ439 and 480 mg PQP. (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  Interventions: Drug: 480 mg Piperaquine phosphate; Drug: 200 mg OZ 439
- Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP (Experimental): 200mg of OZ439 and 640 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  Interventions: Drug: 640 mg Piperaquine phosphate; Drug: 200 mg OZ 439
- Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP (Experimental): 400mg of OZ439 and 480 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  Interventions: Drug: 480 mg Piperaquine phosphate; Drug: 400 mg OZ 439
- Cohort 1Treatment Group D and Cohort 3 Treatment group A : 400mg of OZ439 and 640 mg PQP (Experimental): 400mg of OZ439 and 640 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  Interventions: Drug: 640 mg Piperaquine phosphate; Drug: 400 mg OZ 439
- Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP (Experimental): 800mg of OZ439 and 960 mg PQP.
  Interventions: Drug: 800 mg OZ 439; Drug: 960 mg PQP
- Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP (Experimental): 200mg of OZ439 and 320 mg PQP.
  Interventions: Drug: 400 mg OZ 439; Drug: 320 mg PQP
- Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP (Experimental): 800mg of OZ439 and 640 mg PQP
  Interventions: Drug: 640 mg Piperaquine phosphate; Drug: 800 mg OZ 439

INTERVENTIONS:
Drug: 480 mg Piperaquine phosphate — 480 mg Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  Other Names: PQP
  Arms: Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP; Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP
Drug: 640 mg Piperaquine phosphate — 640 mg Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  Other Names: PQP
  Arms: Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP; Cohort 1Treatment Group D and Cohort 3 Treatment group A : 400mg of OZ439 and 640 mg PQP; Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP
Drug: 200 mg OZ 439 — 200 mg OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension
  Other Names: Artefenomel
  Arms: Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP; Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP
Drug: 400 mg OZ 439 — 400 mg OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension
  Other Names: Artefenomel
  Arms: Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP; Cohort 1Treatment Group D and Cohort 3 Treatment group A : 400mg of OZ439 and 640 mg PQP; Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP
Drug: 800 mg OZ 439 — 800 mg OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension
  Other Names: Artefenomel
  Arms: Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP; Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP
Drug: 960 mg PQP — 960 mg Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  Other Names: Piperaquine Phosphate
  Arms: Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP
Drug: 320 mg PQP — 320 mg Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  Other Names: Piperaquine Phosphate
  Arms: Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP

SUMMARY:
A single-centre Phase 1b study to assess the safety, tolerability, pharmacokinetic profile, and antimalarial activity of single doses of coadministered artefenomel (OZ439) and piperaquine phosphate (PQP) against early Plasmodium falciparum blood stage infection in healthy adult volunteers.

DETAILED DESCRIPTION:
This is a single-centre, open-label, adaptive, study using the P. falciparum induced blood stage malaria (IBSM) inoculum as a model to characterise the pharmacodynamic (PD) activity of combined single dose administration of OZ439 and PQP.

The study will be conducted in a maximum of three cohorts (up to 8 subjects per cohort) using up to 4 different doses of OZ439 and PQP in each cohort. Subjects will be malaria naïve healthy males or females, aged between 18-55 years old, who meet all of the inclusion criteria and none of the exclusion criteria.

The first cohort will be composed of 4 groups of 2 subjects each. Subjects will be randomised into one of 4 dose groups and administered single oral doses of OZ439 and PQP in combination The combined dose of OZ439 and PQP will be different for each of the 4 groups in this cohort as shown in Table 1.

Table 1 OZ439 and PQP Cohort 1 Dose Drug Dose group

1A 1B 1C 1D OZ439 (mg) 200 200 400 400 PQP (mg) 480 640 480 640

The data captured from this first cohort will be used to determine the relationship between OZ439 and PQP concentrations and parasitaemia levels. Based on safety and tolerability data up to Day 35 post-dose, and pharmacokinetic/pharmacodynamic (PK/PD) analysis outcomes (based on PD data up to Day 35 and PK data up to Day 28 post-dose) of the drugs given in combination, the dose(s) for the subsequent cohort will be determined. A similar analysis will be done at the end of cohort 2 combining cohorts 1 and 2 data to decide the dose(s) to be tested in cohort 3. This will be decided by the funding sponsor and the Principal Investigator following review of the data by the Safety and Data Review Team (SDRT) and scientific evaluation.

The doses used in all cohorts will not exceed the maximum acceptable doses predefined for this study (800 mg for OZ439 and 1440 mg for PQP) as determined in previous safety, pilot efficacy and phase 2 studies.

Each subject will be inoculated on Day 0 with approximately 2,800 viable parasites of P. falciparum-infected human erythrocytes administered intravenously. Subjects will be followed up daily via phone call or text message on Days 1 to 3 post-inoculation to solicit any AEs.

Subjects will then come to the clinical unit once daily from Day 4 until presence of asexual parasites is established by quantitative polymerase chain reaction (qPCR) targeting the 18S rRNA gene (referred to hereafter as malaria 18S qPCR). Once qPCR becomes positive and until OZ439 and PQP administration, subjects will come to the clinical unit twice-daily, separated by approximately 12 hours, for clinical evaluation and blood sampling.

Subjects will be admitted to the clinical unit for single dose administration of OZ439 and PQP 8 days after malaria inoculation or at Investigators discretion (i.e. as per parasitaemia levels). Subjects will be followed up as inpatients for at least 72 hours to ensure tolerance of the investigational treatments and clinical response, then if clinically well on an outpatient basis for safety and clearance of malaria parasites via qPCR.

After discharge from the clinical unit, subjects will be followed up regularly for safety assessments, PK sampling, clinical evaluation, and malaria qPCR blood sampling until 35 days after OZ439 and PQP administration. All subjects will receive a standard course of therapy with Riamet® (artemether-lumefantrine) 34 days after OZ439 and PQP administration, or earlier in the event of failure of clearance of parasitaemia or recrudescence of parasitaemia. The presence of gametocytes in subjects' blood will be determined by parasite lifecycle stage qRT-PCR or by the presence of stable low level parasitaemia. If gametocytes are present at the time of treatment with Riamet®, Primacin™ (primaquine) will also be administered as a single oral dose.

AEs (AEs) will be monitored via telephone, within the clinical unit, and on outpatient review after malaria challenge inoculation and antimalarial study drugs administration. Blood samples for safety evaluation, malaria monitoring, and red blood cell antibodies will be drawn at screening and/or baseline and at nominated times after malaria challenge.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (male and female) subjects between 18 and 55 years of age inclusive, who do not live alone (from inoculation day until at least the end of the Riamet® treatment) and will be contactable and available for the duration of the trial and contactable up to 2 weeks following the End of Study visit (approximately 8.5 weeks).
2. Body weight minimum 50 kg, body mass index between 18 and 32 kg/m2, inclusive.
3. Certified as healthy by a comprehensive clinical assessment (detailed medical history, complete physical examination and special investigations).
4. Vital signs after 5 minutes resting in supine position:

   * 90 mmHg ≤ systolic blood pressure (SBP) ≤ 140 mmHg,
   * 40 mmHg ≤ diastolic blood pressure (DBP) ≤ 90 mmHg,
   * 40 bpm ≤ heart rate (HR) ≤ 100 bpm.
5. Must have QTcF ≤450 ms, QTcB ≤450 ms for male subjects, QTcF ≤470 ms, QTcB ≤470 ms for female subjects and PR interval ≤210 ms at screening and at pre-inoculation on inoculation day.
6. Heterosexual women of childbearing potential should be surgically sterile or using an insertable, injectable, transdermal or combination oral contraceptive approved by the TGA combined with a barrier contraceptive for the duration of the study, and have negative results on a urine pregnancy test done before inoculation. Abstinent, heterosexual female subjects must agree to start a double method if they start a sexual relationship during the study. Adequate contraception does not apply to subjects of childbearing potential with same sex partners (abstinence from penile-vaginal intercourse), when this is their preferred and usual lifestyle. Female subjects with same sex partners must not be planning in vitro fertilisation within the required contraception period.

   Women of non-childbearing potential who will not require contraception during the study are defined as: post-menopausal (spontaneous amenorrhoea for ≥ 12 months, or spontaneous amenorrhoea for 6-12 months and follicle-stimulating hormone (FSH) ≥ 40 IU/mL; either should be together with the absence of oral contraceptive use for > 12 months).

   Male subjects participating must agree to use a double-barrier method of contraception including condom plus diaphragm or condom plus intrauterine device or condom plus stable oral/transdermal/injectable hormonal contraceptive by the female partner from the time of informed consent through to 90 days after the last dose of OZ439 and PQP. Abstinent male subjects must agree to start a double-barrier method if they begin sexual relationships during the study and up to 90 days after the last dose of study drug.

   Male subjects with female partners that are surgically sterile, or male subjects who have undergone sterilisation and have had testing to confirm the success of the sterilisation may also be included.
7. Having given written informed consent prior to undertaking any study-related procedure.
8. Must be willing and able to communicate and participate in the whole study. -

Exclusion Criteria:

1. Haematology, clinical chemistry, coagulation or urinalysis results at screening or on admission prior to Inoculation or IMP administration that are outside of Sponsor-approved clinically acceptable laboratory ranges documented in the laboratory manual or are considered clinically relevant.
2. Any history of malaria or participation in a previous malaria challenge study.
3. Must not have travelled to or lived (>2 weeks) in a malaria-endemic region during the past 12 months or planned travel to a malaria-endemic region during the course of the study (for endemic regions see https://map.ox.ac.uk/country-profiles/#!/). Bali is not considered a malaria-endemic region.
4. Participation in any investigational product study within the 12 weeks preceding IMP administration.
5. Has evidence of increased cardiovascular disease risk (defined as >10%, 5-year risk for those greater than 35 years of age, as determined by the Australian Absolute Cardiovascular Disease Risk Calculator (http://www.cvdcheck.org.au/)). Risk factors include sex, age,systolic blood pressure (mm/Hg), smoking status, total and HDL cholesterol (mmol/L), and reported diabetes status.
6. Symptomatic postural hypotension at screening on two consecutive readings, irrespective of the decrease in blood pressure, or asymptomatic postural hypotension defined as a decrease in systolic blood pressure ≥20 mmHg within 2-3 minutes when changing from supine to standing position.
7. History of splenectomy.
8. History or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies (including but not limited to allergy to any of the antimalarial rescue medications to be used in the study), or history of anaphylaxis or other severe allergic reactions. Note. Subjects with seasonal allergies/hay fever, house dust mite or allergy to animals that are untreated and asymptomatic at the time of dosing can be enrolled in the study
9. History of convulsion (including intravenous drug or vaccine-induced episodes) Note. A medical history of a single febrile convulsion during childhood is not an exclusion criterion.
10. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease (HIV or other immuno-deficiencies), insulin-dependent and non-insulin dependent diabetes (excluding glucose intolerance if exclusion criterion 4 is met), progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, porphyria, psoriasis, rheumatoid arthritis, asthma, epilepsy, or obsessive-compulsive disorder.
11. History of malignancy of any organ system (other than localised basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within 5 years of screening, regardless of whether there is evidence of local recurrence or metastases.
12. Subjects with history of schizophrenia, bi-polar disease, or other severe (disabling) chronic psychiatric diagnosis including depression or receiving psychiatric drugs or who has been hospitalised within the past 5 years prior to enrolment for psychiatric illness, history of suicide attempt, or confinement for danger to self or others.
13. History of serious psychiatric condition that may affect participation in the study or preclude compliance with the protocol, including but not limited to past or present psychoses, disorders requiring lithium, a history of attempted or planned suicide, more than one previous episode of major depression, any previous single episode of major depression lasting for or requiring treatment for more than 6 months, or any episode of major depression during the 5 years preceding screening.The Beck Depression Inventory (Appendix 4) will be used as an objective tool for the assessment of depression at screening. In addition to the conditions listed above, subjects with a score of 20 or more on the Beck Depression Inventory and/or a response of 1, 2 or 3 for item 9 of this inventory (related to suicidal ideation) will not be eligible for participation. These subjects will be referred to a general practitioner or medical specialist as appropriate. Subjects with a Beck score of 17 to 19 may be enrolled at the discretion of the Investigator if they do not have a history of the psychiatric conditions mentioned in this criterion and their mental state is not considered to pose additional risk to the health of the subject or to the execution of the study and interpretation of the data gathered.
14. History of recurrent headache (e.g. tension-type, cluster or migraine) with a frequency of ≥2 episodes per month on average and/or severe enough to require medical therapy.
15. Presence of acute infectious disease or fever (e.g. sublingual temperature ≥38.5°C) within the 5 days prior to inoculation with malaria parasites.
16. Evidence of acute illness within the 4 weeks prior to screening that the Investigator deems may compromise subject safety.
17. Significant inter-current disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.
18. Subject has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion (e.g. gastrectomy, diarrhoea).
19. Blood donation of any volume within 1 month before inclusion, or participation in any research study involving blood sampling (more than 450 mL/unit of blood), or blood donation to Australian Red Cross Blood Service (Blood Service) or other blood bank during the 8 weeks prior to the treatment drug dose in the study.
20. Subject unwilling to defer blood donations to the Blood Service for at least 6 months.
21. Medical requirement for intravenous immunoglobulin or blood transfusions.
22. Subject who has ever received a blood transfusion.
23. History or presence of alcohol abuse (alcohol consumption more than 40 g per day) or drug habituation, or any prior intravenous usage of an illicit substance.
24. Tobacco use of more than 5 cigarettes or equivalent per day, and unable to stop smoking for the duration of the clinical unit confinement.
25. Female subject who is breastfeeding.
26. Any vaccination within the last 28 days.
27. Any corticosteroids, anti-inflammatory drugs, immunomodulators or anticoagulants. Any subject currently receiving or having previously received immunosuppressive therapy (including systemic steroids, adrenocorticotrophic hormone or inhaled steroids) at a dose or duration associated with hypothalamic-pituitary-adrenal axis suppression (e.g. 1 mg/kg/day prednisone, chronic use of inhaled high potency corticosteroids such as budesonide 800 μg/day or fluticasone 750 μg, or equivalent).
28. Any recent (<6 weeks) or current systemic therapy with an antibiotic or drug with potential antimalarial activity (e.g. chloroquine, piperaquine phosphate, benzodiazepine, flunarizine, fluoxetine, tetracycline, azithromycin, clindamycin, doxycycline etc.).
29. Ingestion of any poppy seeds within the 24 hours prior to the screening blood test (subjects will be advised by phone not to consume any poppy seeds in this time period).
30. Excessive consumption of beverages or food containing xanthine bases including Red Bull, chocolate, coffee etc. (more than 400 mg caffeine per day, equivalent to more than 4 cups of coffee per day).
31. Unwillingness to abstain from consumption of grapefruit or Seville oranges from inoculation day until end of Riamet® treatment.
32. Unwillingness to abstain from consumption of quinine containing foods/beverages such as tonic water and lemon bitter, from inoculation day until end of Riamet® treatment.
33. Use of prescription drugs or non-prescription drugs or herbal supplements (such as St John's Wort), within 14 days or 5 half-lives (whichever is longer) prior to the malaria inoculation. As an exception, ibuprofen (preferred) may be used at doses of up to 1.2 g/day or paracetamol at doses of up to 4 g/day after discussion with the Investigator. Limited use of other non-prescription medications or dietary supplements, not believed to affect subject safety or the overall results of the study, may be permitted on a case-by-case basis following approval by the Sponsor in consultation with the Investigator. Subjects are requested to refrain from taking non-approved concomitant medications from recruitment until the conclusion of the study.
34. Any subject who, in the judgment of the Investigator, is likely to be non-compliant during the study, or is unable to cooperate because of a language problem or poor mental development.
35. Any subject in the exclusion period of a previous study according to applicable regulations.
36. Any subject who is the Principal Investigator or any sub-Investigator, research assistant, pharmacist, study coordinator, or other staff thereof, directly involved in conducting the study.
37. Any subject without a good peripheral venous access. Biological status
38. Positive result on any of the following tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
39. Positive urine drug test. Any drug listed in Section 7.2.1 in the urine drug screen unless there is an explanation acceptable to the Investigator (e.g., the subject has stated in advance that they consumed a prescription or over-the-counter product which contained the detected drug) and/or the subject has a negative urine drug screen on retest by the pathology laboratory. Any subject testing positive for acetaminophen (paracetamol) at screening may still be eligible for study participation, at the Investigator's discretion.
40. Positive alcohol breath test.
41. Cardiac/QT risk:

    * Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
    * History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
    * Electrolyte disturbances, particularly hypokalaemia, hypocalcaemia, or hypomagnesaemia.
    * ECG abnormalities in the standard 12-lead ECG (at screening or at pre-inoculation on inoculation day) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analyses.
42. Known hypersensitivity to artesunate or any of its excipients, artemether or other artemisinin derivatives, piperaquine phosphate, proguanil/atovaquone, primaquine, or 4-aminoquinolines.

    -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2019-04-19 (Actual); Study Completion 2019-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Webster, Dr, Study Chair — QIMR Berghofer Medical Research Institute
Locations (1):
- Q-Pharm, Herston, Queensland, Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abd-Rahman AN, Kaschek D, Kummel A, Webster R, Potter AJ, Odedra A, Woolley SD, Llewellyn S, Webb L, Marquart L, Chalon S, Gaaloul ME, McCarthy JS, Mohrle JJ, Barber BE. Characterizing the pharmacological interaction of the antimalarial combination artefenomel-piperaquine in healthy volunteers with induced blood-stage Plasmodium falciparum to predict efficacy in patients with malaria. BMC Med. 2024 Nov 28;22(1):563. doi: 10.1186/s12916-024-03787-0. PMID 39609822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: phase 1 unit
Groups:
- Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP: 200mg of OZ439 and 480 mg PQP. (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  480 mg Piperaquine phosphate (PQP): Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  200 mg OZ 439: OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension)
- Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP: 200mg of OZ439 and 640 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  640 mg Piperaquine phosphate (PQP): Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  200 mg OZ 439: OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension)
- Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP: 400mg of OZ439 and 480 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  480 mg Piperaquine phosphate (PQP): Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  400 mg OZ 439: OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension)
- Cohort 1, Group D and Cohort 3 Group A: :Treatment 400mg of OZ439 and 640 mg PQP: 400mg of OZ439 and 640 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  640 mg Piperaquine phosphate (PQP): Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  400 mg OZ 439: OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension)
- Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP: 800mg of OZ439 and 480 mg PQP. (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  960 mg Piperaquine phosphate (PQP): Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  200 mg OZ 439: OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension)
- Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP: 200mg of OZ439 and 480 mg PQP. (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  320 mg Piperaquine phosphate (PQP): Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  200 mg OZ 439: OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension)
- Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP: 800mg of OZ439 and 640 mg PQP. (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  320 mg Piperaquine phosphate (PQP): Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  200 mg OZ 439: OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension)
Period: Overall Study
Arm/Group | Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP | Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP | Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP | Cohort 1, Group D and Cohort 3 Group A: :Treatment 400mg of OZ439 and 640 mg PQP | Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP | Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP | Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP
Started | 2 | 2 | 2 | 6 | 4 | 4 | 4
Completed | 2 | 2 | 2 | 5 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP | Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP | Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP | Cohort 1, Group D and Cohort 3 Group A: :Treatment 400mg of OZ439 and 640 mg PQP | Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP | Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP | Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP | Total
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 4 | 4 | 4 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 6 | 4 | 4 | 4 | 24
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (7.78) | 23.0 (1.41) | 40.5 (17.68) | 23.5 (4.09) | 21.3 (2.22) | 23.8 (3.59) | 20.0 (1.41) | 25.0 (7.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 1 | 6 | 1 | 2 | 2 | 12
  Male | 2 | 2 | 1 | 0 | 3 | 2 | 2 | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 1 | 0 | 2 | 5 | 3 | 4 | 4 | 19
  More than one race | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 2 | 2 | 2 | 6 | 4 | 4 | 4 | 24

OUTCOME MEASURES:

1. Primary Outcome: Characterize the PK/PD Relationship Between OZ439 and PQP Plasma Concentrations (Cmax)
Description: Maximum observed drug concentration in observed individual concentration-time profile.
Time Frame: PK data up to Day 28 post-dose
Population: all patients who were treated with OZ and PQP
Measure: Geometric Mean (Standard Deviation); unit: ng/L
Arm/Group | Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP | Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP | Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP | Cohort 1, Group D and Cohort 3 Group A: :Treatment 400mg of OZ439 and 640 mg PQP | Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP | Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP | Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 4 | 4 | 4
ng/L
  Cmax OZ 439 | 0.2582 (0.05869) | 0.4145 (0.1669) | 0.8829 (0.4108) | 0.6835 (0.2292) | 2.135 (0.7359) | 0.3208 (0.5176) | 1.910 (0.3029)
  Cmax PQP | 0.1168 (0.03599) | 0.05441 (0.02072) | 0.06458 (0.02871) | 0.1048 (0.1081) | 0.4104 (0.07950) | 0.04609 (0.07520) | 0.1860 (0.1489)

2. Primary Outcome: Characterize the PK/PD Relationship Between OZ439 and PQP and Blood Stage Asexual Parasitaemia Measured by Parasite Reduction Ratio at 48 Hours (PRR48)
Description: Ratio between parasitemia at the onset of drug treatment and 48 hours later. The PRR is defined as the ratio of the number of parasites at time of treatment divided by the number after a given amount of time has elapsed post-treatment. This time period is normally 48 hours as this is the time taken for P. falciparum parasites to pass through their asexual erythrocytic life cycle.
Time Frame: From IP administration to 48 hours
Population: all participants who were treated with OZ and PQP
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP | Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP | Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP | Cohort 1, Group D and Cohort 3 Group A: :Treatment 400mg of OZ439 and 640 mg PQP | Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP | Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP | Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 4 | 4 | 4
ratio | 219 [121 to 395] | 151 [100 to 228] | 3777 [1970 to 7243] | 5038 [3340 to 7598] | 9656 [5445 to 17125] | 78 [57 to 109] | 3632 [2289 to 5763]

3. Primary Outcome: Characterize the PK/PD Relationship Between OZ439 and PQP and Blood Stage Asexual Parasitaemia Measured by Parasite Clearance Half-life
Description: PCt1/2 = Parasite Clearance Half-life;
Time Frame: from IP administration to 108 hours
Population: participants
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP | Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP | Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP | Cohort 1, Group D and Cohort 3 Group A: :Treatment 400mg of OZ439 and 640 mg PQP | Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP | Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP | Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP
Number analyzed (Participants) | 2 | 2 | 2 | 6 | 4 | 4 | 4
hours | 6.18 [5.57 to 6.93] | 6.63 [6.13 to 7.22] | 4.04 [3.74 to 4.39] | 3.90 [3.72 to 4.10] | 3.63 [3.41 to 3.87] | 7.63 [7.10 to 8.25] | 4.06 [3.84 to 4.30]

ADVERSE EVENTS:
Time Frame: 38 Days: Treatment Emergent Adverse Events were collected from the time of treatment up to the end of the study.
Groups:
- Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP: 200mg of OZ439 and 640 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  640 mg Piperaquine phosphate: 640 mg Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  200 mg OZ 439: 200 mg OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension
- Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP: 400mg of OZ439 and 480 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  480 mg Piperaquine phosphate: 480 mg Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  400 mg OZ 439: 400 mg OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension
- Cohort 1Treatment Group D and Cohort 3 Treatment Group A : 400mg of OZ439 and 640 mg PQP: 400mg of OZ439 and 640 mg PQP.
  (OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension) and PQP.
  640 mg Piperaquine phosphate: 640 mg Piperaquine is a bis 4-aminoquinoline and was used mainly in China from the 1960's to the 1980's as an antimalarial monotherapy.
  400 mg OZ 439: 400 mg OZ439 + α-tocopherol polyethylene glycol 1000 succinate (TPGS) granules for oral suspension
Arm/Group | Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP | Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP | Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP | Cohort 1Treatment Group D and Cohort 3 Treatment Group A : 400mg of OZ439 and 640 mg PQP | Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP | Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP | Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/6 | 0/4 | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/6 | 0/4 | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 2/2 | 1/2 | 2/2 | 4/6 | 4/4 | 3/4 | 4/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Treatment Group A: 200mg of OZ439 and 480 mg PQP (N=2) | Cohort 1:Treatment Group B: 200mg of OZ439 and 640 mg PQP (N=2) | Cohort 1:Treatment Group C: 400mg of OZ439 and 480 mg PQP (N=2) | Cohort 1Treatment Group D and Cohort 3 Treatment Group A : 400mg of OZ439 and 640 mg PQP (N=6) | Cohort 2: Treatment Group A: 800mg of OZ439 and 960 mg PQP (N=4) | Cohort 2: Treatment Group B: 200mg of OZ439 and 320 mg PQP (N=4) | Cohort 3: Treatment Group B: 800mg of OZ439 and 640 mg PQP (N=4)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Bruise at vessel puncture site (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall in haemoglobin (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fall in lymphocyte count (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall in neutrophil count (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Prolonged QT interval (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising at vascular access site (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-27): https://cdn.clinicaltrials.gov/large-docs/49/NCT03542149/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-29): https://cdn.clinicaltrials.gov/large-docs/49/NCT03542149/SAP_001.pdf